CLINICAL TRIAL: NCT04098692
Title: A Phase 1, Two-part, Open-label, Single-oral-dose Study to Investigate the Absolute Bioavailability and Absorption, Pharmacokinetics, Distribution, Metabolism, and Excretion of [14C]-Derazantinib in Healthy Male Subjects
Brief Title: Mass Balance and Pharmacokinetics Study of Derazantinib in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DZB-CS-102
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — derazantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm: Derazantinib (Part 1 and Part 2) (Experimental): * Part 1: 300 mg Derazantinib oral administration followed by 100 μg [14C]-Derazantinib intravenous microdose
  * Part 2: 300 mg [14C]-Derazantinib oral administration
  Interventions: Drug: Derazantinib capsule; Drug: [14C]-Derazantinib solution for infusion; Drug: [14C]-Derazantinib capsule

INTERVENTIONS:
Drug: Derazantinib capsule — 300 mg derazantinib oral administration (3x100 mg capsules)
Drug: [14C]-Derazantinib solution for infusion — 100 μg [14C]-derazantinib intravenous administration
Drug: [14C]-Derazantinib capsule — 300 mg [14C]-derazantinib oral administration (3x100 mg capsules)

SUMMARY:
This is a Phase 1, two-part, open-label, single centre, single arm study in healthy male subjects to investigate the oral PK, intravenous (IV) PK, mass balance, bioavailability and metabolites profiling and identification of derazantinib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age 18 to ≤ 55 years (Part 1)
* Age 30 to ≤ 65 years (Part 2)
* Body mass index of 18.0 to 29.0 kg/m² and a minimum body weight of 50 kg
* Must have regular bowel movements
* Must agree to adhere to the contraception requirements

Exclusion Criteria:

* Male subjects with pregnant partners
* Subjects who have received any investigational medicine in a clinical research study within the previous 3 months
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* History of any drug or alcohol abuse in the 12 months prior to dosing
* Regular alcohol consumption in males > 21 units per week
* Smokers and users of e-cigarettes and nicotine replacement products and those who have used these products within the last 3 months
* Radiation exposure (diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
* Participation in any study involving administration of any [14C]-labelled compound within 12 months prior to screening (Part 1 only)
* Excessive caffeine consumption within 14 days prior to screening, defined as 800 mg per day (approximately 6 large cups of coffee)
* Subjects who do not have suitable veins
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the Investigator
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results, or history of immunodeficiency diseases, including a positive HIV (ELISA and western blot) test result
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of < 70 mL/min using the Cockcroft-Gault equation
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder or current clinical evidence of any corneal or retinal disorder
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
* Known hypersensitivity or allergy to natural rubber latex
* History of any food allergies
* History of clinically significant ECG abnormalities
* Familial history of sick-sinus syndrome
* Recent (within the last 3 years) and/or recurrent history of autonomic dysfunction
* Recent (within the last 3 years) and/or recurrent history of acute or chronic bronchospastic disease (including asthma disease, treated or not treated)
* History of malignancy of any organ system (other than localised basal cell carcinoma of the skin), treated or untreated, within the past 5 years
* Use of any prescription drugs (including vaccines), herbal supplements (such as St. John's Wort, homeopathic preparations), within 4 weeks prior to initial dosing, and/or over-the-counter medication, dietary supplements (vitamins and minerals included) within 2 weeks prior to initial dosing
* Donation or loss of 400 mL or more of blood and/or plasma within 3 months prior to initial dosing
* Any history or presence of frequent episodes of diarrhoea (defined as an increase of 4 to 6 stools per day over usual individual defecation pattern).
* Significant illness within 2 weeks prior to initial dosing
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardise the subject in case of participation in the study.

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Assessment of the PK of total radioactivity, [14C]-derazantinib, derazantinib, and BAL0122840: Cmax | up to Day 50
  Assessment of the maximum observed plasma concentration (Cmax)
Assessment of the PK of total radioactivity, [14C]-derazantinib, derazantinib, and BAL0122840: Tmax | up to Day 50
  Assessment of the time from dosing at which Cmax was apparent (Tmax)
Assessment of the PK of total radioactivity, [14C]-derazantinib, derazantinib, and BAL0122840: t½ | up to Day 50
  Assessment of the apparent terminal elimination half-life (t½)
Assessment of the PK of total radioactivity, [14C]-derazantinib, derazantinib, and BAL0122840: AUC0-t | up to Day 50
  Assessment of the area under the concentration-time curve from dosing to the last measurable concentration (AUC0-t)
Assessment of the PK of total radioactivity, [14C]-derazantinib, derazantinib, and BAL0122840: AUC0-inf | up to Day 50
  Assessment of the area under the concentration-time curve from dosing extrapolated to infinity (AUC0-inf)
Assessment of the PK of total radioactivity, [14C]-derazantinib, derazantinib, and BAL0122840: Tlast | up to Day 50
  Assessment of the time of the last measurable (positive) concentration (Tlast)
Assessment of the PK of [14C]-derazantinib: CL | up to Day 50
  Assessment of the total clearance (CL)
Assessment of the PK of [14C]-derazantinib: Vss | up to Day 50
  Assessment of the volume of distribution at steady state (Vss)
Assessment of the PK of [14C]-derazantinib: Vd | up to Day 50
  Assessment of the volume of distribution (Vd)
Assessment of the PK of derazantinib: CL/F | up to Day 50
  Apparent total clearance (CL/F)
Assessment of the PK of derazantinib: F | up to Day 50
  Absolute bioavailability (F)
Assessment of the rate and routes of excretion, and the mass balance of total radioactivity in urine and faeces and in all excreta | up to Day 50
  Assessment of total radioactivity by measuring the amount excreted (Ae), Ae as a percentage of the administered dose (%Ae), cumulative recovery (CumAe), and cumulative recovery expressed as a percentage of the dose (Cum%Ae)

CONTACTS AND LOCATIONS:
Overall Officials: Nand Singh, MD, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom